CLINICAL TRIAL: NCT07406243
Title: Mitochondrial-Targeted Antioxidant Supplementation for Improving Cerebrovascular Function in Postmenopausal Women
Brief Title: Oral Antioxidant Therapy Targeted to the Mitochondria for Improving Brain Artery Health in Postmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7559; K01HL177339 (NIH)
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Aging; Postmenopause
MeSH Terms: interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MitoQ, 20 mg/day (Experimental): Each MitoQ capsule contains 20 mg of mitoquinol mesylate. Dosage: 20 mg orally per day for 3 months.
  Interventions: Dietary Supplement: Mitoquinone (MitoQ)
- Placebo (Placebo Comparator): Matched placebo capsules.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mitoquinone (MitoQ) — MitoQ is a biochemically modified form of ubiquinol
  Other Names:
  Mitoquinol
  Arms: MitoQ, 20 mg/day
Dietary Supplement: Placebo — Each placebo capsule contains inert excipient and is identical in appearance
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if 3 months of taking the dietary supplement MitoQ [a mitochondria-targeted antioxidant that targets to reduce mitochondrial reactive oxygen species (mitoROS)] works to treat age- and menopause-related reductions in brain artery (cerebrovascular) function in postmenopausal women 60 years of age or older free of clinical disease. The main questions it aims to answer are:

Does MitoQ improve cerebrovascular function in postmenopausal women?

If so, does MitoQ improve cerebrovascular function by lowering mitoROS in these arteries?

Researchers will compare MitoQ to a placebo (a look-alike substance that contains no drug) to see if MitoQ can improve cerebrovascular function by lowering mitoROS in arteries involved in brain health and function.

Participants will:

Take MitoQ (20 mg/day) or a placebo every day for 3 months

Visit the research laboratory at baseline and then after 3 months for cerebrovascular testing; there is also a check-in visit at 6 weeks, which is the halfway point

Keep track of symptoms and events during their treatment period to report to the study team

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older;
* Postmenopausal women defined as at least 1 year without menses as self-reported;
* Estrogen-deficient; no hormone therapies (e.g., estrogen, progesterone, testosterone, DHEA, oral contraceptives, etc.) within the previous 6 months;
* Ability to provide informed consent;
* Willing to accept random assignment to condition;
* Body mass index (BMI) ≤35 kg/m2;
* Mini-mental state examination score ≥21;
* Weight stable in the prior 3 months;
* Abstinence from antioxidant or CoQ10 therapy for 3 months; and
* Absence of clinical disease as determined by the physician of record following a medical history and blood chemistries

Exclusion Criteria:

* History of uncontrolled hypertension;
* Currently meeting aerobic exercise guidelines of ≥75 mins/week of vigorous or ≥150 mins/week of moderate intensity exercise as assessed by Modified Activity Questionnaire;
* Current smoker;
* Alcohol dependence or abuse;
* Other chronic medical conditions; and
* Subject report of blood donation within 8 weeks prior to enrolling.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in cerebrovascular conductance at 3 months | 3 months
  Middle cerebral artery blood velocity in response to hypercapnia normalized for changes in end-tidal carbon dioxide and blood pressure

SECONDARY OUTCOMES:
Change from baseline in cerebrovascular reactivity at 3 months | 3 months
  Middle cerebral artery blood velocity in response to hypercapnia normalized to changes in end-tidal carbon dioxide
Change from baseline in mitochondrial oxidative stress-mediated suppression of cerebrovascular conductance at 3 months | 3 months
  Cerebrovascular conductance to hypercapnia following administration of a supratherapeutic dose of MitoQ (160 mg) known to scavenge mitochondrial reactive oxygen species
Change from baseline in mitochondrial oxidative stress-mediated suppression of cerebrovascular reactivity at 3 months | 3 months
  Cerebrovascular reactviity to hypercapnia following administration of a supratherapeutic dose of MitoQ (160 mg) known to scavenge mitochondrial reactive oxygen species
Change from baseline in internal carotid artery dilation in response to hypercapnia at 3 months | 3 months
  Cerebrovascular endothelium-dependent dilation
Change from baseline in mitochondrial oxidative stress-mediated suppression of internal carotid artery dilation at 3 months | 3 months
  Internal carotid artery dilation to hypercapnia following administration of a supratherapeutic dose of MitoQ (160 mg) known to scavenge mitochondrial reactive oxygen species
Change from baseline in total cerebral blood flow at 3 months | 3 months
  The amount of blood flow feeding the brain at rest
Change from baseline in cerebrovascular stiffness at 3 months | 3 months
  Resting middle cerebral artery pulsatility index
Change from baseline in carotid artery compliance at 3 months | 3 months
  Change in diameter of carotid artery for a given change in pressure
Change from baseline in mitochondrial oxidative stress-mediated suppression of carotid artery compliance at 3 months | 3 months
  Carotid artery compliance following administration of a supratherapeutic dose of MitoQ (160 mg) known to scavenge mitochondrial reactive oxygen specie

OTHER OUTCOMES:
Change from baseline in serum exposure-induced arterial endothelial function at 3 months | 3 months
  Donor mouse arterial endothelium-dependent dilation after treatment with serum from subjects
Change from baseline in serum exposure-induced arterial stiffness at 3 months | 3 months
  Donor mouse arterial elastic modulus after treatment with serum from subjects
Change from baseline in circulating oxidized low-density lipoprotein at 3 months | 3 months
  Blood marker of oxidative stress

CONTACTS AND LOCATIONS:
Locations (1):
- Translational Physiology Laboratory within the Food Science Clinical Research Laboratory, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD will not be on a publicly available repository, however, any or all data may be made available upon reasonable request and collaboration.
Supporting Information: Study Protocol
Time Frame: We will publish a study protocol paper within the first year of the study to enhance rigor and reproducibility of trial.
Access Criteria: Those seeking access to the data with a research question and open for collaboration will be considered.